CLINICAL TRIAL: NCT01126190
Title: A Randomized, Double-Blind, Active Comparator, Non-Inferiority Study of Subcutaneously Administered Neugranin (Recombinant Human Albumin-Human Granulocyte Colony Stimulating Factor) or Pegfilgrastim in Subjects With Breast Cancer Receiving Myelosuppressive Chemotherapy (Doxorubicin/Docetaxel), Followed by a Single-Arm, Open-Label Phase of Subcutaneously Administered Neugranin
Brief Title: Neugranin in Breast Cancer Participants Receiving Doxorubicin/Docetaxel
Acronym: NEUGR-003
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NEUGR-003
Record Dates: First submitted 2010-05-04; First posted 2010-05-19 (Estimated); Results first posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-02

CONDITIONS: Chemotherapy-induced Neutropenia
MeSH Terms: interventions — balugrastim; pegfilgrastim; Drug Therapy; Doxorubicin; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Double-Blind Phase: Pegfilgrastim (Active Comparator): Participants will receive pegfilgrastim 6 milligrams (mg), administered by subcutaneous (SC) injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days). The chemotherapy regimen consists of doxorubicin 60 mg/square meter (m^2) and docetaxel 75 mg/m^2 administered sequentially by intravenous (IV) infusion on Day 1 of treatment for up to four 21-day cycles.
  Interventions: Biological: Pegfilgrastim; Drug: Chemotherapy
- Double-Blind Phase: Neugranin 40 mg (Experimental): Participants will receive neugranin 40 mg, administered by SC injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days). The chemotherapy regimen consists of doxorubicin 60 mg/m^2 and docetaxel 75 mg/m^2 administered sequentially by IV infusion on Day 1 of treatment for up to four 21-day cycles.
  Interventions: Biological: Neugranin; Drug: Chemotherapy
- Open-Label Phase: Neugranin 40 mg (Experimental): Participants will receive neugranin 40 mg, administered by SC injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days). The chemotherapy regimen consists of doxorubicin 60 mg/m^2 and docetaxel 75 mg/m^2 administered sequentially by IV infusion on Day 1 of treatment for up to four 21-day cycles.
  Interventions: Biological: Neugranin; Drug: Chemotherapy

INTERVENTIONS:
Biological: Neugranin — Neugranin will be administered per dose and schedule specified in the arm description.
  Other Names: Balugrastim
  Arms: Double-Blind Phase: Neugranin 40 mg; Open-Label Phase: Neugranin 40 mg
Biological: Pegfilgrastim — Pegfilgrastim will be administered per dose and schedule specified in the arm description.
  Other Names: Neulasta
  Arms: Double-Blind Phase: Pegfilgrastim
Drug: Chemotherapy — The chemotherapy regimen for this trial consists of doxorubicin 60 mg/m^2 and docetaxel 75 mg/m^2 in combination
  Other Names: Doxorubicin/Docetaxel

SUMMARY:
Determination of the effect of neugranin on the duration and severity of severe neutropenia in participants receiving doxorubicin in combination with docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer participants scheduled to receive the AT regimen (doxorubicin/ docetaxel)

Exclusion Criteria:

* Participants may have received no more than 1 prior chemotherapy regimen (including adjuvant therapy if given within the last 12 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2010-06-30 (Actual); Primary Completion 2012-02-29 (Actual); Study Completion 2012-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (59):
- Bulgaria (8):
  - Teva Investigational Site 3502, Gabrovo
  - Teva Investigational Site 3511, Plovdiv
  - Teva Investigational Site 3504, Rousse
  - Teva Investigational Site 3501, Shumen
  - Teva Investigational Site 3506, Sofia District
  - Teva Investigational Site 3503, Stara Zagora
  - Teva Investigational Site 3505, Varna
  - Teva Investigational Site 3507, Veliko Tarnovo
- Romania (8):
  - Teva Investigational Site 4001, Baia Mare, Maramures County
  - Teva Investigational Site 4009, Brasov
  - Teva Investigational Site 4004, Bucharest
  - Teva Investigational Site 4002, Cluj-Napoca
  - Teva Investigational Site 4011, Cluj-Napoca
  - Teva Investigational Site 4005, Craiova, Dolj County
  - Teva Investigational Site 4010, Lasi County
  - Teva Investigational Site 4007, Timișoara
- Russia (23):
  - Teva Investigational Site 0714, Arkhangelsk
  - Teva Investigational Site 0707, Chelyabinsk
  - Teva Investigational Site 0708, Ivanovo
  - Teva Investigational Site 0721, Kazan'
  - Teva Investigational Site 0709, Krasnodar
  - Teva Investigational Site 0711, Kursk
  - Teva Investigational Site 0713, Leningrad Region
  - Teva Investigational Site 0710, Moscow
  - Teva Investigational Site 0703, Moscow
  - Teva Investigational Site 0716, Nizhny Novgorod
  - Teva Investigational Site 0720, Oryol
  - Teva Investigational Site 0724, Pyatigorsk
  - Teva Investigational Site 0725, Rostov-on-Don
  - Teva Investigational Site 0704, Saint Petersburg
  - Teva Investigational Site 0722, Saint Petersburg
  - Teva Investigational Site 0706, Saint Petersburg
  - Teva Investigational Site 0715, Saint Petersburg
  - Teva Investigational Site 0712, Samara
  - Teva Investigational Site 0723, Sochi
  - Teva Investigational Site 0717, Tambov
  - Teva Investigational Site 0719, Ufa
  - Teva Investigational Site 0705, Yaroslavl
  - Teva Investigational Site 0702, Yekaterinburg
- Serbia (4):
  - Teva Investigational Site 8102, Belgrade
  - Teva Investigational Site 8103, Belgrade
  - Teva Investigational Site 8104, Kragujevac
  - Teva Investigational Site 8105, Niš
- Ukraine (16):
  - Teva Investigational Site 3807, Chernihiv
  - Teva Investigational Site 3805, Chernivtsi
  - Teva Investigational Site 3802, Dnipropetrovsk
  - Teva Investigational Site 3811, Donetsk
  - Teva Investigational Site 3806, Ivano-Frankivsk
  - Teva Investigational Site 3814, Kharkiv
  - Teva Investigational Site 3804, Kharkiv
  - Teva Investigational Site 3816, Kharkiv
  - Teva Investigational Site 3803, Khmelnytskyi
  - Teva Investigational Site 3808, Kyiv
  - Teva Investigational Site 3817, Kyiv
  - Teva Investigational Site 3812, Lviv
  - Teva Investigational Site 3809, Mariupol, Donetsk Region
  - Teva Investigational Site 3801, Odesa
  - Teva Investigational Site 3815, Sumy
  - Teva Investigational Site 3810, Uzhhorod

REFERENCES:
- [Derived] Volovat C, Gladkov OA, Bondarenko IM, Barash S, Buchner A, Bias P, Adar L, Avisar N. Efficacy and safety of balugrastim compared with pegfilgrastim in patients with breast cancer receiving chemotherapy. Clin Breast Cancer. 2014 Apr;14(2):101-8. doi: 10.1016/j.clbc.2013.10.001. Epub 2013 Oct 25. PMID 24485296

RESULTS

PARTICIPANT FLOW:
Groups:
- Double-Blind Phase: Pegfilgrastim: Participants received pegfilgrastim 6 milligrams (mg), administered by subcutaneous (SC) injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days). The chemotherapy regimen consisted of doxorubicin 60 mg/square meter (m^2) and docetaxel 75 mg/m^2 administered sequentially by intravenous (IV) infusion on Day 1 of treatment for up to four 21-day cycles.
- Double-Blind Phase: Neugranin 40 mg; Open-Label Phase: Neugranin 40 mg: Participants received neugranin 40 mg, administered by SC injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days). The chemotherapy regimen consisted of doxorubicin 60 mg/m^2 and docetaxel 75 mg/m^2 administered sequentially by IV infusion on Day 1 of treatment for up to four 21-day cycles.
Period: Double-Blind Phase
Arm/Group | Double-Blind Phase: Pegfilgrastim | Double-Blind Phase: Neugranin 40 mg | Open-Label Phase: Neugranin 40 mg
Started | 151 | 153 | 0
Received at Least 1 Dose of Study Drug | 150 | 153 | 0
Completed Without a Major Protocol Deviation | 148 | 150 | 77
Completed | 145 | 138 | 0
Not Completed | 6 | 15 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 5 | 0
Not completed — Request of Investigator | 1 | 0 | 0
Not completed — Treatment Failure/Disease Progression | 0 | 4 | 0
Not completed — Non-compliance | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 3 | 0
Period: Open-Label Phase
Arm/Group | Double-Blind Phase: Pegfilgrastim | Double-Blind Phase: Neugranin 40 mg | Open-Label Phase: Neugranin 40 mg
Started | 0 | 0 | 77
Received at Least 1 Dose of Study Drug | 0 | 0 | 77
Completed | 0 | 0 | 66
Not Completed | 0 | 0 | 11
Not completed — Death | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Population: For the double-blind period, the intent-to-treat (ITT) population included all randomized participants. For the open-label period, the ITT population included all enrolled participants who satisfied eligibility criteria.
Groups:
- Double-Blind Phase: Pegfilgrastim: Participants received pegfilgrastim 6 mg, administered by SC injection once per chemotherapy cycle (approximately 24 hours after chemotherapy administration) for up to 4 cycles (each cycle length = 21 days). The chemotherapy regimen consisted of doxorubicin 60 mg/m^2 and docetaxel 75 mg/m^2 administered sequentially by IV infusion on Day 1 of treatment for up to four 21-day cycles.
- Total: Total of all reporting groups
Arm/Group | Double-Blind Phase: Pegfilgrastim | Double-Blind Phase: Neugranin 40 mg | Open-Label Phase: Neugranin 40 mg | Total
Number analyzed (Participants) | 151 | 153 | 77 | 381
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (9.65) | 51.5 (10.28) | 52.2 (10.22) | 51.4 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 153 | 77 | 381
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 151 | 153 | 77 | 381
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Double-Blind Phase: Duration of Severe Neutropenia in Cycle 1
Description: Severe neutropenia was defined as Grade 4 neutropenia (absolute neutrophil count [ANC] <0.5 x 10^9/liter [L]). The duration of severe neutropenia was calculated by cycle as the number of days from the first day in which the ANC fell below 0.5 x 10^9/L after beginning a chemotherapy cycle until the participant had an ANC ≥0.5 x 10^9/L within the cycle.
Time Frame: Cycle 1 (cycle length = 21 days)
Population: Per protocol (PP) population included all data from randomized participants that were obtained prior to experiencing major protocol violations.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Double-Blind Phase: Pegfilgrastim | Double-Blind Phase: Neugranin 40 mg
Number analyzed (Participants) | 148 | 150
days | 1.0 (1.08) | 1.1 (1.13)
Statistical Analysis 1: Comparison: Double-Blind Phase: Pegfilgrastim vs Double-Blind Phase: Neugranin 40 mg; For the primary non-inferiority endpoint of cycle 1 DSN, the 95% confidence interval (CI) for difference in DSN was calculated by stratified bootstrap resampling; Test type: Non-Inferiority — Non-inferiority was demonstrated if the upper endpoint of the CI for the difference in mean DSN was less than or equal to 0.62 days; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.13 to 0.37]

2. Secondary Outcome: Double-Blind Phase: Number of Participants With Febrile Neutropenia
Description: Febrile neutropenia was defined as an imputed or observed ANC <0.5 x 10^9/L and body temperature >38.5 degrees celsius (°C) occurring on the same day and for more than one hour (axillary measurement). Number of participants with febrile neutropenia over all cycles (Cycles 1 to 4) has been reported.
Time Frame: Cycles 1-4 (each cycle = 21 days)
Population: PP population included all data from randomized participants that were obtained prior to experiencing major protocol violations.
Measure: Number; unit: participants
Arm/Group | Double-Blind Phase: Pegfilgrastim | Double-Blind Phase: Neugranin 40 mg
Number analyzed (Participants) | 148 | 150
participants | 4 | 2

3. Primary Outcome: Open-Label Phase: Duration of Severe Neutropenia in Cycle 1
Description: Severe neutropenia was defined as Grade 4 neutropenia (ANC <0.5 x 10^9/L). The duration of severe neutropenia was calculated by cycle as the number of days from the first day in which the ANC fell below 0.5 x 10^9/L after beginning a chemotherapy cycle until the participant had an ANC ≥0.5 x 10^9/L within the cycle. There was no planned statistical analysis for the open-label phase arm.
Time Frame: Cycle 1 (cycle length = 21 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Open-Label Phase: Neugranin 40 mg
Number analyzed (Participants) | 77
days | 1.0 (1.03)

4. Secondary Outcome: Open-Label Phase: Number of Participants With Febrile Neutropenia
Description: Febrile neutropenia was defined as an imputed or observed ANC <0.5 x 10^9/L and body temperature >38.5 °C occurring on the same day and for more than one hour (axillary measurement). Number of participants with febrile neutropenia over all cycles (Cycles 1 to 4) has been reported.
Time Frame: Cycles 1-4 (each cycle = 21 days)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Open-Label Phase: Neugranin 40 mg
Number analyzed (Participants) | 77
participants | 2

ADVERSE EVENTS:
Time Frame: From the start of study drug administration through 30 days following the final dose of study drug (up to 114 days)
Description: For the double-blind period, the safety population included all randomized participants who received at least 1 dose of randomized study drug.
  For the open-label period, the safety population included all participants who received at least 1 dose of neugranin.
Arm/Group | Double-Blind Phase: Pegfilgrastim | Double-Blind Phase: Neugranin 40 mg | Open-Label Phase: Neugranin 40 mg
All-Cause Mortality (participants affected / at risk) | 0/150 | 2/153 | 2/77
Serious Adverse Events (participants affected / at risk) | 7/150 | 6/153 | 6/77
Other Adverse Events (participants affected / at risk) | 134/150 | 139/153 | 71/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Phase: Pegfilgrastim (N=150) | Double-Blind Phase: Neugranin 40 mg (N=153) | Open-Label Phase: Neugranin 40 mg (N=77)
Agranulocytosis (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cyanosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular complication associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Subdiaphragmatic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Phase: Pegfilgrastim (N=150) | Double-Blind Phase: Neugranin 40 mg (N=153) | Open-Label Phase: Neugranin 40 mg (N=77)
Anaemia (Blood and lymphatic system disorders) | 10 (34) | 12 (68) | 5 (6)
Leukopenia (Blood and lymphatic system disorders) | 22 (73) | 26 (92) | 19 (63)
Neutropenia (Blood and lymphatic system disorders) | 40 (176) | 45 (164) | 16 (46)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (33) | 21 (60) | 2 (4)
Vertigo (Ear and labyrinth disorders) | 7 (11) | 6 (8) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 17 (24) | 22 (34) | 8 (9)
Nausea (Gastrointestinal disorders) | 62 (146) | 56 (144) | 26 (56)
Stomatitis (Gastrointestinal disorders) | 9 (12) | 11 (15) | 3 (7)
Vomiting (Gastrointestinal disorders) | 15 (18) | 16 (26) | 5 (5)
Asthenia (General disorders) | 33 (79) | 42 (107) | 22 (48)
Fatigue (General disorders) | 15 (31) | 16 (35) | 6 (10)
Decreased appetite (Metabolism and nutrition disorders) | 20 (46) | 24 (54) | 10 (16)
Bone pain (Musculoskeletal and connective tissue disorders) | 16 (26) | 18 (29) | 14 (39)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 10 (17) | 7 (10)
Headache (Nervous system disorders) | 16 (23) | 20 (33) | 7 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 114 (135) | 124 (153) | 60 (76)
Erythema (Skin and subcutaneous tissue disorders) | 12 (28) | 12 (28) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.